CLINICAL TRIAL: NCT03777410
Title: Mass Accumulation Rate (MAR) as a Predictive Biomarker in Multiple Myeloma
Status: Terminated | Type: Observational
Why Stopped: Insufficient pace of enrollment due to changes in MM SOC practices
Sponsor: Travera Inc (Industry)
Collaborators: Dana-Farber Cancer Institute (Other); Massachusetts General Hospital (Other); Weill Medical College of Cornell University (Other); City of Hope Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: TRV-001
Record Dates: First submitted 2018-12-14; First posted 2018-12-17 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Multiple Myeloma in Relapse
Keywords: functional; biomarker; multiple myeloma; phenotypic; biophysical
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Vanguard: (CLOSED TO ENROLLMENT) Bone marrow (BM) from this cohort of up to 30 treatment naïve subjects with a diagnosis of multiple myeloma (MM) will first be used to define sample processing pipeline performance and optimal drug dosages before sites on the study proceed to mass accumulation rate (MAR) testing of BM from the relapsed/refractory MM (RRMM) subject cohort.
- Relapsed/Refractory MM: BM from this cohort of 100 relapsed subjects with a diagnosis of MM will be used to test the MAR assay's accuracy of condition by matching conditions tested in vitro to the patient's planned course of therapy. This is the main study cohort described in the Eligibility section.

SUMMARY:
This study will collect bone marrow (BM) aspirate samples from patients with relapsed refractory multiple myeloma (RRMM) prior to the start of a new treatment regimen for the purposes of prospectively measuring single-cell mass accumulation rate (MAR) as a biomarker of patient response to that regimen.

The primary study objective is to explore whether the single-cell MAR biomarker can predict patient response in RRMM patients. In order to enable this primary objective, two patient cohorts will be required. First, a small vanguard cohort of patients with treatment naïve disease to define drug concentrations used for testing, and second, the main RRMM patient cohort. Data will be collected to estimate the biomarker's predictive properties (accuracy, sensitivity, specificity), and to support improvement of the MAR biomarker through additional research and discovery within the study dataset.

ELIGIBILITY:
Inclusion Criteria:

1. Written Informed Consent provided by patient
2. MM, with the following conditions:

(CLOSED) *For patients in the Vanguard cohort*

1. Treatment naïve disease with BM clinically indicated

*For patients in the RRMM cohort*

1. Relapsed/refractory disease with BM samples clinically indicated
2. Within 4-weeks prior to initiation of 2nd-line or later therapy
3. Patient's oncologist must be planning to change the patient's next line of treatment to a monotherapy or combination therapy composed exclusively of drugs from the following list: Bortezomib (Velcade), Carfilzomib (Kyprolis), Lenalidomide (Revlimid), Pomalidomide (Pomalyst), Cyclophosphamide (Cytoxan), Dexamethasone, Ixazomib (Ninlaro), Venetoclax (Venclexta), Selinexor (Xpovio)

Exclusion Criteria:

1. Unable or unwilling to provide informed consent
2. Daratumumab/Elotuzumab or other antibody-based therapeutic regimens as immediately planned treatment (as prior therapy is acceptable)
3. Patient enrolled/enrolling in a clinical trial where data or specimen sharing provisions preclude use in this study
4. Prior exposure to CAR-T therapy
5. Prior allogeneic stem cell transplant
6. Has received any systemic chemotherapy or RT, including palliative, within 7 days prior to BM biopsy
7. Has received any Ab therapy within 4 weeks prior to BM biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient's pursuing initial care for their multiple myeloma at one of the 6 study sites
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Best Response 4 months | 0-4 months
  The best International Myeloma Working Group (IMWG) response of each patient over 4 months of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Nikhil C Munshi, M.D., Principal Investigator — Dana-Farber Cancer Institute; Cara Rosenbaum, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (4):
- United States (4):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Weill Cornell Medicine - New York Presbyterian, New York, New York

IPD SHARING:
Plan to Share IPD: No